CLINICAL TRIAL: NCT06444152
Title: Prevalence of Epstein-Barr Virus Infection in HIV Infected and HIV Uninfected Patients Presenting With Lymphomas in Botswana
Brief Title: Prevalence of Epstein-Barr Virus Infection
Status: Active, not recruiting | Type: Observational
Sponsor: University of Pennsylvania (Other)
Collaborators: University of Botswana (Other)
Responsible Party: Sponsor
Other Study IDs: 831640
Record Dates: First submitted 2024-05-29; First posted 2024-06-05 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Lymph Node Excision Biopsy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Sample analysis — This study is analyzing stored samples

SUMMARY:
This will be a cross sectional, pilot study to determine the burden of EBV related lymphomas in this population. Patient information including demographics and HIV status, history of HIV infection, HIV viral load and CD4 counts and ART history will be retrieved from the integrated patient management system (IPMS) Lymph node excision biopsy samples, collected at NHL between 2012 and 2017, from the patient with a diagnosis of lymphoma will be retrieved using IPMS from National Health Laboratory and analyzed by immunohistochemistry.

DETAILED DESCRIPTION:
Lymph node excision biopsy samples,which have been formalin fixed and paraffin embedded, of 50 HIV-infected and 50 HIV-uninfected patients from the patient with a diagnosis of lymphoma, will be retrieved using IPMS from National Health Laboratory. Archived diagnostic biopsy material will be collected from NHL between 2012 and 2017 (5 years). They will be analyzed by immunohistochemistry using LMP-1/EBNA1/ENNA2 staining, either alone or combined which indicates a diagnosis of EBV infection.

We will compute rates of EBV associated lymphomas among HIV infected and HIV uninfected individuals using descriptive statistics. The students t-test will be used for continuous variables while the Pearson's chi squared test (or Fisher's exact test where appropriate) will be used to compare categorical variables. Significance will be assigned for P values of 0.05 or less

ELIGIBILITY:
Inclusion Criteria:

* All available lymph node biopsy samples with a diagnosis of lymphoma and complete data of HIV status, HIV viral load and CD4 counts and ART history will be retrieved from IPMS.

Exclusion Criteria:

* Samples with incomplete data

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Formalin fixed paraffin embedded tissue (FFPE) of lymph node excision biopsy samples from the patient with a diagnosis of lymphoma
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2023-08-01 (Actual); Primary Completion 2027-12-20 (Estimated); Study Completion 2027-12-20 (Estimated)

PRIMARY OUTCOMES:
Burden of EBV | 12 months
  The prevalence of EBV associated lymphomas among HIV-infected and HIV-uninfected patients in excision biopsy specimens of lymph nodes. This will be a cross sectional, pilot study to determine the burden of EBV related lymphomas in this population.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Botswana, Gaborone, Botswana

IPD SHARING:
Plan to Share IPD: No